CLINICAL TRIAL: NCT00555581
Title: Phase IIA Study of the Safety and Tolerability of the Use of Imatinib Mesylate (Gleevec) in the Treatment of Systemic Sclerosis
Brief Title: Imatinib Mesylate (Gleevec) in the Treatment of Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27049
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Systemic Sclerosis
Keywords: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 400 mg daily of Imatinib Mesylate (Experimental): All patients were treated with imatinib mesylate at a target dose of 400 mg daily by mouth for 12 months. Dose modifications and interruptions were made for AE and were recorded. After 12 months of treatment, imatinib was stopped for 3 months. Patients were reassessed and offered entrance to an extension phase of the trial.
  Interventions: Drug: Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib Mesylate — In initial phase, patients will be treated with Gleevec 400 mg daily for 12 months. In the extension phase, patients will be treated with Gleevec 400 mg daily for 27 months.

SUMMARY:
The purpose of this study is to assess the safety and tolerability of imatinib mesylate (Gleevec) in patients with systemic sclerosis (scleroderma). Gleevec is a medication already FDA approved for the treatment of chronic myelogenous leukemia (CML), gastrointestinal stromal tumors (GIST), dermatofibrosarcoma protuberans tumors, Philadelphia chromosome-positive acute lymphoblastic leukemia, hypereosinophilic syndrome, and aggressive systemic mastocytosis. In-vitro studies have suggested that imatinib may inhibit collagen production by scleroderma fibroblasts, and in mouse models of fibrosis imatinib has been shown to decrease skin thickness.

This is a Phase IIa, single center, prospective open label clinical trial of Gleevec in patients with systemic sclerosis. All patients will be treated with active drug for 12 months. The primary objective of this study will be to determine the safety and tolerability of Gleevec in patients with systemic sclerosis, but important secondary outcomes of relevance will be improvement in disease status as defined by skin scores and indices of pulmonary function.

Patients who complete the initial phase (described above) of the study will be eligible to participate in an extension phase. The purpose of the extension phase of the study is to give patients who participated in the phase IIa clinical trial of Gleevec at the Hospital for Special Surgery the opportunity to continue Gleevec treatment if both the treating physicians and the patient are in agreement that Gleevec had acceptable safety and tolerability, as well as possible efficacy during the initial year of therapy.

DETAILED DESCRIPTION:
Further description of extension phase:

Patients will first be evaluated for inclusion in the extension phase of the study at either the follow-up visit following three month withdrawal from Gleevec treatment or at the visit after the follow-up visit. Patients can undergo evaluation for inclusion in the extension phase up to six months following their completion of the initial one year trial. All patients evaluated for inclusion in the extension phase will sign a new informed consent form detailing the purpose and procedures associated with the extension phase at the initial visit. After the initial visit, patients who meet inclusion criteria will be required to undergo evaluation every three months for the 27 months following initiation of treatment, or more frequently if deemed clinically necessary. Treatment will consist of Gleevec, at doses ranging from 100 to 400 mg daily (100 mg pills will be distributed for oral administration). At each study visit, a history and physical exam will be performed and urine and blood tests will be conducted for disease activity and organ function. Additional blood for research may also be collected at study visits. The Modified Rodnan Skin Score will be measured to assess the degree of skin involvement associated with the patient's disease. Patients will also continue to complete questionnaires about their ability to function and quality of life.

Patients will be financially responsible for all professional and clinical services, as well as all laboratory and diagnostic tests, associated with the extension phase of the study. All co-pays, deductibles and co-insurances will be paid by the participants. Any additional costs for parking and travel the patients incur as a result of participating in the extension phase will not be reimbursed by the study. Novartis Pharmaceuticals will donate drug supply.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to eighteen years.
2. Clinical diagnosis of diffuse systemic sclerosis by ACR criteria, with a stable modified Rodnan skin score in the one month preceding introduction of oral Gleevec therapy. The modified Rodnan skin score must be greater than or equal to sixteen at screening and initiation of therapy.
3. Disease duration of less than or equal to 10 years.
4. Estimated ejection fraction of greater than 50% by echocardiography

Exclusion Criteria:

1. Inability to render informed consent in accordance with institutional guidelines.
2. Disease duration of greater than 10 years.
3. Patients with mixed connective tissue disease or "overlap" (i.e. those who satisfy more than one set of ACR criteria for a rheumatic disease.)
4. Ongoing treatment with other immunosuppressive therapies including cyclophosphamide, azathioprine, mycophenolic acid, methotrexate, or cyclosporine, or use of those medications within 3 months of trial entry.
5. Concurrent serious medical condition which in the opinion of the investigator makes the patient inappropriate for this study such as uncontrollable CHF, arrhythmia, severe pulmonary or systemic hypertension, severe GI involvement, serum creatinine of greater than 2.0, active infection, severe diabetes, unstable atherosclerotic cardiovascular disease, malignancy, HIV, or severe peripheral vascular disease.
6. The use of other anti-fibrotic agents including colchicine, D-penicillamine, minocycline, or Type 1 oral Collagen in the three months prior to enrollment.
7. Limited scleroderma.
8. Systemic sclerosis-like illness associated with environmental or ingested agents such as toxic rapeseed oil, vinyl chloride, or bleomycin.
9. A positive pregnancy at entry into this study. Men and women with reproductive potential will be required to use effective means of contraception through the course of the study.
10. Use in the prior month of corticosteroids at doses exceeding the equivalent of prednisone 10 mg daily. Use of corticosteroid at < 10 mg of prednisone can continue but not be increased during the course of the study.
11. Participation in another clinical research study involving the evaluation of another investigational drug within ninety days of entry into this study.
12. The presence of severe lung disease as defined by a diffusion capacity of less than 30% of predicted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Spiera, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Derived] Haddon DJ, Wand HE, Jarrell JA, Spiera RF, Utz PJ, Gordon JK, Chung LS. Proteomic Analysis of Sera from Individuals with Diffuse Cutaneous Systemic Sclerosis Reveals a Multianalyte Signature Associated with Clinical Improvement during Imatinib Mesylate Treatment. J Rheumatol. 2017 May;44(5):631-638. doi: 10.3899/jrheum.160833. Epub 2017 Mar 15. PMID 28298564
- [Derived] Spiera RF, Gordon JK, Mersten JN, Magro CM, Mehta M, Wildman HF, Kloiber S, Kirou KA, Lyman S, Crow MK. Imatinib mesylate (Gleevec) in the treatment of diffuse cutaneous systemic sclerosis: results of a 1-year, phase IIa, single-arm, open-label clinical trial. Ann Rheum Dis. 2011 Jun;70(6):1003-9. doi: 10.1136/ard.2010.143974. Epub 2011 Mar 11. PMID 21398330
- See also: Clinical Trials - HSS — http://www.hss.edu/clinical-trials_gleevec-sclerosis-scleroderma.asp
- See also: Related Info — http://www.hss.edu/clinical-trials.asp

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 400 mg Daily of Imatinib Mesylate
Started | 30
Completed | 24
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | 400 mg Daily of Imatinib Mesylate
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 48 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Disease Duration [Mean (Standard Deviation); unit: years]
  Early | 2.1 (1.2)
  Late | 6.1 (1.6)
Anti-Scl70 positive [Count of Participants; unit: Participants] | 9
MRSS at baseline [Mean (Standard Deviation); unit: units on a scale] — The Modified Rodnan Skin Score (MRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. In each of these areas, the skin score is evaluated by manual palpation. The skin score is 0 for uninvolved skin, 1 for mild thickening, 2 for moderate thickening, and 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas. The minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease.
  units on a scale | 30.3 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Improvement in the Modified Rodnan Skin Score
Description: Improvement in the Modified Rodnan Skin Score (MRSS) is measured by Mean change (and 95% Confidence Interval) from Baseline mean to Month 12 mean.Measure Description: The Modified Rodnan Skin Score (MRSS) measures dermal skin thickness through the examination of 17 body areas: fingers, hands, forearms, arms, feet, legs, and thighs (in pairs), and face, chest, and abdomen. The skin score is 0 for uninvolved skin through 3 for severe thickening (hidebound skin). The total skin score is the sum of the skin scores of the individual areas. The minimum score is 0 and the maximum score is 51. A higher score indicates greater severity of disease. The mean change in MRSS represents the average change in total skin score from baseline to month 12.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 400 mg Daily of Imatinib Mesylate
Number analyzed (Participants) | 24
units on a scale | -6.6 [-8.7 to -4.5]

2. Secondary Outcome: Improvement in Indices of Pulmonary Function Measured by Change in FVC % Predicted
Description: This outcome measure includes patients with and without the presence of Interstitial Lung Disease (ILD). Forced vital capacity (FVC) is the amount of air that can be forcibly exhaled from the lungs after taking a deep breath. It is used to determine the severity of lung disease. Improvement in FVC % predicted is measured by Mean change (and 95% Confidence Interval) from Baseline mean to Month 12 mean. Results are compared to the predicted values that are calculated from a patients age, size, weight, and sex. Results are considered normal if FVC is 80 percent or more of the predicted value. Mean change in FVC % predicted is measured by the average change in FVC% percent predicted from baseline to month 12.
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: FVC%
Arm/Group | 400 mg Daily of Imatinib Mesylate
Number analyzed (Participants) | 22
FVC% | 6.4 [1.9 to 10.9]

3. Secondary Outcome: Improvement in Indices of Pulmonary Function Measured by Change DLCO hb Adj % Predicted
Description: This outcome measure includes patients with and without the presence of Interstitial Lung Disease (ILD). Diffusion capacity of the lungs for carbon monoxide (DLCO) measures how much oxygen travels from the alveoli of the lungs to the blood stream. DLCO is adjusted for hemoglobin as small changes in hemoglobin concentration can affect the carbon monoxide transfer. DLCO results are compared to normal values for a patient's height, age, sex, and ethnicity. A DLCO result that is at least 80% of the predicted value is considered normal. Improvement in DLCO hb adj % predicted is measured by Mean change (and 95% Confidence Interval) from Baseline mean to Month 12 mean (the average change in DLCO hb adj% from baseline to month 12).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: DLCO%
Arm/Group | 400 mg Daily of Imatinib Mesylate
Number analyzed (Participants) | 22
DLCO% | 5.5 [-1.5 to 12.4]

4. Secondary Outcome: Change From Baseline at Month 12 in Short Form-36 (SF-36) Questionnaire:Mental Component Summary
Description: The Short Form 36 (SF-36) is a validated 36 item questionnaire which measures quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health. The mental component score is composed of a subset of the 8 health domains. Each component is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 is equivalent to no disability.The SF-36 mental component can be obtained by looking at the mean average of all the emotionally relevant items. Change in Short Form 36 mental (SF-36 MC) is measured by Mean change (and 95 % Confidence Interval) from Baseline mean to Month 12 mean (the average change in SF-36 mental component from baseline to month 12).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 400 mg Daily of Imatinib Mesylate
Number analyzed (Participants) | 24
units on a scale | -6.6 [-12.5 to -0.7]

5. Secondary Outcome: Scleroderma Health Assessment Questionnaire Disability Index
Description: The Scleroderma Health Assessment Questionnaire (SHAQ) consist of the Health Assessment Questionnaire (HAQ) and 8 other domains which include scales looking at pain, patient global assessment, vascular, digital ulcers, lung involvement, and gastrointestinal involvement. It addresses scleroderma related manifestations that contribute to disability. It is a quality of life measure. Each question is scored from 0 (without difficulty) to 3 (unable to do). Some domains in the SHAQ are visual analog scales that are measured first and then changed to a 0-3 scale.
  The maximum from each category is added together and divided by the number of categories completed. Change in Scleroderma Health Assessment Questionnaire Disability Index (SHAQ-DI) is measured as Mean Change (and 95% Confidence Interval) from Baseline mean to Month 12 mean (the average change in SHAQ-DI from baseline to month 12).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 400 mg Daily of Imatinib Mesylate
Number analyzed (Participants) | 24
units on a scale | 0.02 [-0.15 to 0.18]

6. Secondary Outcome: Change From Baseline at Month 12 in Short Form-36 (SF-36) Questionnaire: Physical Component Summary
Description: The Short Form 36 (SF-36) is a 36 item questionnaire which measures quality of life across eight domains: physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, general health. The physical component score is composed of a subset of the 8 health domains.The SF-36 physical component can be obtained by looking at the mean average of all the physically relevant items. Each component is directly transformed into a 0 to 100 scale on the assumption that each question carries equal weight. A score of 0 is equal to maximum disability, and a score of 100 is equivalent to no disability. Change in Short Form 36 physical component (SF-36 PC) is measured by Mean change (and 95 % Confidence Interval) from Baseline mean to Month 12 mean (the average change in SF-36 physical component from baseline to month 12).
Time Frame: 12 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | 400 mg Daily of Imatinib Mesylate
Number analyzed (Participants) | 24
units on a scale | 6.8 [1.7 to 15.3]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | 400 mg Daily of Imatinib Mesylate
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 25/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mg Daily of Imatinib Mesylate (N=30)
Haematuria (hospitalisations) (Renal and urinary disorders) | 1 (7)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
C difficile infection (Infections and infestations) | 1 (2)
Infected ulcer (Infections and infestations) | 2 (2)
Death (pneumonia) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute gastroenteritis (Gastrointestinal disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Anaemia Blood Transfusion (Surgical and medical procedures) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fluid Overload (Blood and lymphatic system disorders) | 1 (1)
Rectal proplapse, haemorrhoidal bleed (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Partial small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Bleeding post renal biopsy (hospitalisation) (Surgical and medical procedures) | 1 (1)
Tachyarrhythmia/cardiomyopathy (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 400 mg Daily of Imatinib Mesylate (N=30)
Edema (General disorders) | 25 (33)
Nausea (Metabolism and nutrition disorders) | 22 (22)
Myalgias (Musculoskeletal and connective tissue disorders) | 21 (21)
CK elevation (Blood and lymphatic system disorders) | 13 (13)
Fatigue (General disorders) | 18 (18)
Pyrosis (Gastrointestinal disorders) | 7 (7)
Vomiting (Metabolism and nutrition disorders) | 7 (7)
Weight Loss (Metabolism and nutrition disorders) | 5 (5)
Headaches (Nervous system disorders) | 7 (7)
Effusions (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Erectile Dysfunction (Reproductive system and breast disorders) | 2 (2)
Generalised weakness (General disorders) | 5 (5)
Light-headedness (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No